CLINICAL TRIAL: NCT01564849
Title: The Clinical Efficacy of Topical Nasal Pomegranate Fruit Extract (PFE) for Patients With Chronic Rhinitis, Chronic Sinusitis With or Without Nasal Polyps
Brief Title: The Clinical Efficacy of Topical Nasal Pomegranate Fruit Extract for Patients With Chronic Rhinosinusitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Gan shmuel Group (Other)
Responsible Party: Principal Investigator, Itzhak Braverman, Head Otolarungology Head and Neck Surgery Unit, Hillel Yaffe Medical Center
Other Study IDs: 89-2011
Record Dates: First submitted 2012-03-25; First posted 2012-03-28 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Rhinitis; Sinusitis; Nasal Polyps
Keywords: Pomegranate fruit extract; Sinusitis; rhinitis; nasal polyps
MeSH Terms: conditions — Rhinitis; Sinusitis; Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- chronic rhinitis,
- chronic sinusitis
- nasal polyps
- control rhinitis
- control sinusitis
- control polyps

SUMMARY:
An explosion of interest in the numerous therapeutic properties of Punica granatum over the last decade has led to numerous in vitro, animal, and clinical trials. Pomegranate is a potent antioxidant, superior to red wine and equal to or better than green tea. In addition, anticarcinogenic and anti-inflammatory properties suggest its possible use as a therapy or adjunct for prevention and treatment of several types of cancer and cardiovascular disease. Because of pomegranate's antimicrobial properties, it may aid in preventing infection by dental pathogens, pathogenic E. coli O157:H7, and antibiotic-resistant organisms such as methicillin-resistant Staphylococcus aureus (MRSA) Pomegranate's effect on bacterial pathogens has only been tested in vitro, however, necessitating human trials to refute or substantiate any clinical effect.

The possibility that pomegranate extracts may also have an effect on several other disease processes, such as Alzheimer's and obesity, underscores the need for more clinical research. Currently, numerous clinical trials are in progress exploring the therapeutic potential of pomegranate extracts.

Aim The investigators want to evaluate the effect of Punica granatum components on Chronic sinusitis, nasal polyps and chronic rhinitis.

DETAILED DESCRIPTION:
There are many publications indexed by Medline dealing with pomegranate and Punica granatum and there is interest in pomegranate as a medicinal and nutritional product.

The pomegranate tree, Punica granatum, especially its fruit, possesses a vast ethnomedical history and represents a phytochemical reservoir of heuristic medicinal value. The tree/fruit can be divided into several anatomical compartments: (1) seed,(2) juice, (3) peel, (4) leaf, (5) flower, (6) bark, and (7) roots, each of which has interesting pharmacologic activity. Juice and peels, for example,possess potent antioxidant properties, while juice, peel and oil are all weakly estrogenic and heuristically of interest for the treatment of menopausal symptoms and sequelae. The use of juice, peel and oil have also been shown to possess anticancer activities, including interference with tumor cell proliferation, cell cycle, invasion and angiogenesis. These may be associated with plant based anti-inflammatory effects. The phytochemistry and pharmacological actions of all Punica granatum components suggest a wide range of clinical applications for the treatment and prevention of chronic inflammation.

Pomegranate as few medical applications as gastrointestinal infections, oral wounds and others. There is a publication on the positive use of pomegranate, in reducing of trigeminal pain post Herpes Zoster infection (1). Another work described the synergistic effect of pomegranate extraction and antibiotics for Staphyloccocus Areus (2). Pomegranate extraction was used for viral delay of HIV I in AIDS patients (3).

It's antiviral effect was examined against HSV and RSV (6). There was a positive effect on H7 -E. COLI 0157(4). Pomegranate extraction was found to help as antibacterial effect as other Mexican extraction drugs, for Gastrointestinal infections (5). High concentrations of phenol substances was evaluated in wound healing and it was efficient (7). Methanolic substances from pomegranate extraction was evaluated and found efficient for all the bacteria that was examined (8). Recently pomegranate extraction was found active in antibacterial effect and in synergism with tetracyclin against staphyloccocus Areus with Methicillin resistance (MRSA).

Pomegranate polyphenol extract (PPE) has anti-influenza properties. Using real time PCR, plaque assay, and TCID 50% hemagglutination assay, the investigators have shown that PPE suppresses replication of influenza A virus in MDCK cells. PPE inhibits agglutination of chicken red blood cells (cRBC) by influenza virus and is virucidal. The single-cycle growth conditions indicated that independent of the virucidal effect PPE also inhibits viral RNA replication. PPE did not alter virus ribonucleoprotein (RNP) entry into nucleus or translocation of virus RNP from nucleus to cytoplasm in MDCK cells. The investigators evaluated four major Polyphenols in PPE (ellagic acid, caffeic acid, luteolin, and punicalagin) and demonstrated that punicalagin is the effective, anti-influenza component of PPE. Punicalagin blocked replication of the virus RNA, inhibited agglutination of chicken RBC's by the virus and had virucidal effects. Furthermore, the combination of PPE and oseltamivir synergistically increased the anti-influenza effect of oseltamivir. In conclusion, PPE inhibited the replication of human influenza A/Hong Kong (H3N2) in vitro. Pomegranate extracts should be further studied for therapeutic and prophylactic potential especially for influenza epidemics and pandemics.

Commonly found in many plants, ellagic acid exhibits powerful anticarcinogenic and antioxidant properties, propelling it to the forefront of pomegranate research. Many commercially available pomegranate extracts are being standardized to contain 40-percent (or more) ellagic acid. Lansky's research confirms the synergistic action of several pomegranate constituents is superior to ellagic acid in suppressing prostate cancer. To quote Lansky, "The recent profusion onto the nutraceuticals marketplace of products standardized to 40 percent (or even higher) ellagic acid represents a cynical, lucre-driven attempt to replace the power of the pomegranate with the power of ellagic acid. The pomegranate needs no such tricks or enhancements. It is rather an extraordinary, albeit mysterious (and messy), fruit with a complete medicinal power contained within its juice, peel, and seeds.

Topical applications of pomegranate preparations have been found to be particularly effective for controlling oral inflammation, as well as bacteria and fungal counts in periodontal disease and Candida-associated denture stomatitis. A hydroalcoholic extract of Punica granatum fruit (HAEP) was investigated for antibacterial effect on dental plaque microorganisms. Sixty healthy patients (33 females/27 males; ages 9-25) with fixed orthodontic appliances were randomized to three groups of 20:

(1) control group who rinsed with 15 mL distilled water; (2) a group who rinsed with 15 mL chlorhexidine, a standard antiplaque mouth rinse; and (3) a group who rinsed with a 15-mL HAEP solution. HAEP decreased the number of colony forming units (CFU) of dental plaque bacteria 84 percent, comparable to chlorhexidine (79-percent inhibition) but significantly better than the control rinse (11-percent inhibition). Both HAEP and chlorhexidine were effective against Staphylococcus, Streptococcus, Klebsiella, and Proteus species, as well as E. coli. The ellagitannin, punicalagin, is thought to be the fraction responsible for pomegranate's antibacterial activity.

Bacterial Infections The only human trials examining the antibacterial properties of pomegranate extracts have focused on oral bacteria. However, several in vitro assays demonstrate its bacteriocidal activity against several highly pathogenic and sometimes antibiotic-resistant organisms. Brazilian researchers evaluated the synergistic effect of a P. granatum methanolic extract with five antibiotics on 30 clinical isolates of methicillin-resistant Staphylococcus aureus (MRSA) and methicillin-sensitive S. aureus.75 Antibiotics tested were chloramphenicol, gentamicin, ampicillin, tetracycline, and oxacillin. Although synergistic activity between the pomegranate extract and all five antibiotics was noted in the S. aureus isolates, synergy with ampicillin was the most pronounced. Based on earlier research and the results of this study, the ellagitannin, punicalagin, is thought to be the primary constituent responsible for the observed antibacterial effects. Another organism that can cause significant disease in humans is enterohemorrhagic Escherichia coli (E. coli O157:H7). An ethanolic PPE, one of the two most effective extracts against E. coli O157:H7, was shown to be both bacteriostatic and bacteriocidal, indicating PPE may be an effective adjunct treatment for E. coli O157:H7 infection.

On the above information the investigators will try and evaluate the clinical efficacy of topical nasal Pomegranate fruit extract (PFE) (Punica Granatum) for patients with Chronic rhinitis, chronic sinusitis, nasal polyps and chronic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* above age 18
* under age 80
* patients with chronic rhinitis, sinusitis and nasal polyps
* patients candidates for surgery or medical therapy

Exclusion Criteria:

* Patients that had nasal surgery before
* smokers
* Diabetes, chemotherapy or radiation therapy
* Allergy to yeasts or pomegranate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults suffering from chronic rhinitis, sinusitis and nasal polyps
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2012-04; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Pob 169, Israel